CLINICAL TRIAL: NCT04430192
Title: Study of the Dosimetry, Safety and Potential Benefit of 177Lu-PSMA-617 Radionuclide Therapy Prior to Radical Prostatectomy in Men With High-risk Localised Prostate Cancer
Brief Title: Dosimetry, Safety and Potential Benefit of 177Lu-PSMA-617 Prior to Prostatectomy
Acronym: LuTectomy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: Movember Foundation (Other); Medical Research Future Fund (Other); Endocyte (Industry); E.J. Whitten Foundation Prostate Cancer Research Centre (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19_245
Record Dates: First submitted 2020-05-21; First posted 2020-06-12 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Prostatic Neoplasms
Keywords: 177Lu-PSMA; Prostate Cancer; Radionuclide Therapy; Theranostics; prostate specific membrane antigen
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 177Lu-PSMA-617 followed by prostatectomy (Experimental): 177Lu-PSMA-617 followed by prostatectomy
  Interventions: Drug: 177Lu-PSMA-617

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — Patients 1-10 will be given 5GBq of 177Lu-PSMA. Patients 11-20 will be given 2 cycles of 5GBq of 177Lu-PSMA, separated by 6 weeks.
  Other Names: 177Lu-PSMA; [177Lu]Lu-PSMA-617; Lu-PSMA

SUMMARY:
This clinical trial will evaluate the dosimetry, efficacy and toxicity of Lu-PSMA in men with high PSMA-expressing high-risk localized or locoregional advanced prostate cancer (HRCaP) undergoing radical prostatectomy (RP) and pelvic lymph node dissection (PLND)

DETAILED DESCRIPTION:
This open label, phase I/II non-randomised clinical trial will evaluate the dosimetry, efficacy and toxicity of Lu-PSMA in men with high PSMA-expressing high-risk localized or locoregional advanced prostate cancer (HRCaP) undergoing radical prostatectomy (RP) and pelvic lymph node dissection (PLND). Patients will receive one or two cycles of 177Lu-PSMA followed by surgery. The primary objective is to determine the radiation absorbed dose in the prostate and involved lymph nodes. Secondary objectives include evaluating imaging response to therapy using PSMA-PET, biochemical response, pathological response, adverse effects of Lu-PSMA and surgical safety, and health-related Quality of Life (QoL).

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided written informed consent.
* Male patient aged 18 or over at the time of screening
* Histologically confirmed adenocarcinoma of the prostate, in a patient scheduled for RP and PLND with curative intent
* High or high-intermediate risk localised or locoregional prostate cancer (HRCaP) by European Association of Urology (EAU) criteria, including any of the following:

  * PSA > 20 ng/mL
  * ISUP grade group 3-5
  * Clinical T-stage by digital rectal examination (DRE) of T2c or higher
  * N1 disease (involvement of lymph nodes at or below the bifurcation of the common iliac arteries)
  * defined radiologically (CT/ MRI, or PSMA PET).
* High PSMA avidity on 68Ga-PSMA PET/CT, defined as an SUVmax of ≥ 20
* Normal baseline haematological function; haemoglobin 13.5-17.5g/dl), total white blood cell count (4-11 x 109/l), platelets (150-400 x 109/l), neutrophils (2-7.5 x 109/l) and lymphocytes (1-4 x 109/l)
* Normal baseline serum biochemistry; sodium 135-145 nmol/l, potassium 3.5-5 nmol/l, chloride 98-108 nmol/l, urea 3-9.2 nmol/l, creatinine 60-120μmol/l
* Willing and able to comply with all study requirements including all treatments and required assessments including follow up

Exclusion Criteria:

* Prostate cancer with significant neuroendocrine or other rare variant pathology
* Prior treatment for prostate cancer including radiotherapy and/or androgen deprivation therapy.
* Evidence of metastatic disease involving bone, viscera, or lymph nodes superior to the common iliac bifurcation based on CT, MRI, WBBS or PSMA PET/CT.
* Renal impairment [GFR < 60mL/min].
* Sjogren's syndrome.
* A history of or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
To determine the radiation absorbed dose in the prostate and involved lymph nodes following one or two administrations of Lu-PSMA in men with HRCaP prior to radical prostatectomy | Determined using imaging at 4, 24 and 96 hrs after administration of Lu-PSMA
  Establishing the absorbed radiation dose in the prostate and involved lymph nodes (Gy)

SECONDARY OUTCOMES:
To evaluate the imaging response to therapy using PSMA-PET | 6 weeks following final administration of Lu-PSMA
  PSMA PET response to therapy (complete metabolic response, partial metabolic response, stable metabolic disease, progressive metabolic disease)
To evaluate the biochemical response to therapy | 6 weeks following final administration of Lu-PSMA
  PSA response
To evaluate pathologic response in the prostate following prostatectomy | After prostatectomy, approximately 6 weeks from final Lu-PSMA administration
  Pathological response (complete response, minimal residual disease)
To evaluate toxicity of Lu-PSMA | Until 8 weeks after prostatectomy
  Assessment of toxicity of Lu-PSMA using Common Terminology Criteria for Adverse Events (CTCAE) v5
To evaluate the surgical safety of prostatectomy following Lu-PSMA | Until 8 weeks after prostatectomy
  Surgical safety will be assessed using using the Clavien-Dindo classification of surgical complications
To evaluate overall health-related Quality of Life (QoL) | baseline, immediately before 2nd cycle Lu-PSMA, immediately before surgery, 8 weeks post surgery, annually up to 3 years
  QoL indices will be scored using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire
To evaluate prostate cancer health-related Quality of Life (QoL) | baseline, immediately before 2nd cycle Lu-PSMA, immediately before surgery, 8 weeks post surgery, annually up to 3 years
  QoL indices will be scored using European Organisation for Research and Treatment of Cancer (EORTC) QLQ-PR25 questionnaire
To evaluate patient function and bother after prostatectomy | baseline, immediately before 2nd cycle Lu-PSMA, immediately before surgery, 8 weeks post surgery, annually up to 3 years
  Indices will be scored using the Expanded Prostate Cancer Index Composite (EPIC)-26 questionnaire

OTHER OUTCOMES:
To determine the time to biochemical recurrence (BCR) [PSA>0.2 ng/mL post-RP] | To be determined as it is an exploratory endpoint up to 3 years
  Biochemical recurrence (BCR) will be measured from the time of surgery to the first rise of the PSA to ≥0.2 ng/mL
To determine the relationship between PSMA PET imaging parameters and absorbed dose | baseline PSMA PET within 45 days of Lu-PSMA administration
  Determination of the relationship between screening PSMA PET imaging parameters including molecular tumour volume parameters and absorbed dose in the prostate and involved lymph nodes
To identify tissue and blood and serum biomarkers associated with clinical outcomes | To be determined as it is an exploratory endpoint up to 3 years
  Determination of relevant predictive biomarkers associated with treatment outcomes and response

CONTACTS AND LOCATIONS:
Overall Officials: Declan Murphy, Principal Investigator — Peter MacCallum Cancer Centre, Australia; Michael S Hofman, Principal Investigator — Peter MacCallum Cancer Centre, Australia; John Violet, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Eapen RS, Buteau JP, Jackson P, Mitchell C, Oon SF, Alghazo O, McIntosh L, Dhiantravan N, Scalzo MJ, O'Brien J, Sandhu S, Azad AA, Williams SG, Sharma G, Haskali MB, Bressel M, Chen K, Jenjitranant P, McVey A, Moon D, Lawrentschuk N, Neeson PJ, Murphy DG, Hofman MS. Administering [177Lu]Lu-PSMA-617 Prior to Radical Prostatectomy in Men with High-risk Localised Prostate Cancer (LuTectomy): A Single-centre, Single-arm, Phase 1/2 Study. Eur Urol. 2024 Mar;85(3):217-226. doi: 10.1016/j.eururo.2023.08.026. Epub 2023 Oct 26. PMID 37891072